CLINICAL TRIAL: NCT02170064
Title: Pharmacokinetics, Efficacy and Tolerability of BIA 2-093 in Children and Adolescents With Refractory Partial Epilepsy
Brief Title: Pharmacokinetics, Efficacy and Tolerability of BIA 2-093
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIA-2093-202
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Results first posted 2014-09-01 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-08

CONDITIONS: Epilepsy
Keywords: Epilepsy; BIA 2-093
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (2-6 yrs) (Experimental): At the end of the baseline phase, patients meeting the final selection criteria were admitted to three consecutive 4-week treatment periods in which they received Eslicarbazepine acetate once-daily at the following dosage regimens: 5 mg/kg/day in the first 4 weeks, 15 mg/kg/day in weeks 5-8 and 30 mg/kg/day or 1800 mg/day, whichever less, in weeks 9-12. After the last treatment period, dose was down-titrated during a 2-week period or patient continued receiving Eslicarbazepine acetate ("compassionate use") if both parent(s)/guardian(s)/patient and his/her physician agreed this was in the best patient's interest.
  For Group 1 (2-6 years), oral suspension 50 mg/mL was used. The dose was to be rounded to the nearest 25 mg unit.
  Interventions: Drug: BIA 2-093 (Eslicarbazepine acetate)
- Group 2 (7-11 years) (Experimental): At the end of the baseline phase, patients meeting the final selection criteria were admitted to three consecutive 4-week treatment periods in which they received Eslicarbazepine acetate once-daily at the following dosage regimens: 5 mg/kg/day in the first 4 weeks, 15 mg/kg/day in weeks 5-8 and 30 mg/kg/day or 1800 mg/day, whichever less, in weeks 9-12. After the last treatment period, dose was down-titrated during a 2-week period or patient continued receiving Eslicarbazepine acetate ("compassionate use") if both parent(s)/guardian(s)/patient and his/her physician agreed this was in the best patient's interest.
  For Group 2 (7-11 years) and Group 3 (12-17 years), Eslicarbazepine acetate strengths 200 mg, 400 mg, 600 mg and 800 mg tablets might be used. The dose was to be rounded to the nearest 100 mg unit. Half tablets might be used for dosage adjustment (tablets were scored).
  Interventions: Drug: BIA 2-093 (Eslicarbazepine acetate)
- Group 3 (12-17 years) (Experimental): At the end of the baseline phase, patients meeting the final selection criteria were admitted to three consecutive 4-week treatment periods in which they received Eslicarbazepine acetate once-daily at the following dosage regimens: 5 mg/kg/day in the first 4 weeks, 15 mg/kg/day in weeks 5-8 and 30 mg/kg/day or 1800 mg/day, whichever less, in weeks 9-12. After the last treatment period, dose was down-titrated during a 2-week period or patient continued receiving Eslicarbazepine acetate ("compassionate use") if both parent(s)/guardian(s)/patient and his/her physician agreed this was in the best patient's interest.
  For Group 2 (7-11 years) and Group 3 (12-17 years), Eslicarbazepine acetate strengths 200 mg, 400 mg, 600 mg and 800 mg tablets might be used. The dose was to be rounded to the nearest 100 mg unit. Half tablets might be used for dosage adjustment (tablets were scored).
  Interventions: Drug: BIA 2-093 (Eslicarbazepine acetate)

INTERVENTIONS:
Drug: BIA 2-093 (Eslicarbazepine acetate) — Eslicarbazepine acetate administered at increasing daily doses of 5 mg/kg, 15 mg/kg, and 30 mg/kg (or 1800 mg, whichever less); once-daily; oral route

SUMMARY:
The purpose of this study is to characterize the pharmacokinetics of Eslicarbazepine acetate in children and adolescents with epilepsy.

DETAILED DESCRIPTION:
This clinical study was planned to be performed as an open-label, single-centre, multiple-dose study, in 30 paediatric epileptic patients distributed by 3 age groups of 10 patients each: 2-6 years [Group 1], 7-11 years [Group 2], and 12-17 years [Group 3].

The study was constituted by a 4-week baseline phase, followed by 3 consecutive 4-week treatment periods with Eslicarbazepine acetate in which patients received Eslicarbazepine acetate once-daily at the following dosage regimens: 5 mg/kg/day (weeks 1-4), 15 mg/kg/day (weeks 5-8) and 30 mg/kg/day or 1800 mg/day, whichever less (weeks 9-12). At the end of each 4-week treatment period, patients were hospitalised and serial blood samples for drug assays were obtained over a dosing interval.

After the last treatment period or in the event of premature discontinuation, the dose had to be down-titrated during a 2-week period. After the last treatment period patient could continue receiving Eslicarbazepine acetate ("compassionate use") if both parent(s)/guardian(s) /patient and his/her physician agreed this was in the best patient's interest. A follow-up visit occurred approximately 4 weeks after the last hospitalisation or early discontinuation.

ELIGIBILITY:
Inclusion Criteria:

The following inclusion criteria were applied in selecting patients for participation in the trial.

Patient was eligible for entry into the baseline phase if he/she fulfilled the following criteria at Visit 1:

* Written informed consent given by the parent(s)/guardian(s), and by the patient when appropriate.
* Male or female patient aged between 2 and 17 years.
* Body weight within the 10th and 90th percentiles, by age and sex.
* A documented diagnosis of partial-onset seizures (simple or complex seizures with or without secondary generalisation), classified according to the International Classification of Epileptic Seizures.
* Currently treated with 1 to 3 AEDs (any except OXC or CBZ), in a stable dosage regimen during at least 1 month prior to screening.
* Good general health (apart from epilepsy) based on medical history and physical examination.
* In case of a female patient, she was premenarchal, surgically sterile or presented a urine pregnancy test consistent with a non-gravid state and practiced an effective non-hormonal contraception method.

At Visit 2, patient was eligible for entry into the Eslicarbazepine acetate treatment phase if he/she fulfilled the following criteria:

* At least 4 partial-onset seizures during the last 4 weeks of the baseline phase.
* Brain CT scan or MRI that excluded rapidly progressive neurological diseases.
* ECG without clinically significant abnormalities.
* Good general health (apart from epilepsy) based on medical history, physical examination and laboratory tests at screening.
* Diaries satisfactorily completed by the patient or his/her caregiver during the baseline phase.
* Satisfactory compliance with the study requirements during the baseline phase.
* In case of a female patient of childbearing potential, she presented a urine pregnancy test consistent with a non-gravid state and practiced an effective non-hormonal contraception method.

Exclusion Criteria:

Patient was not allowed for entry into the screening phase if he/she fulfilled the following criteria at Visit 1:

* Primarily generalised epilepsy.
* Clinically relevant medical condition, other than epilepsy.
* History of status epilepticus in the last 3 months.
* History of suicide attempt.
* History of alcohol or drug abuse.
* History of hypersensitivity or intolerance to OXC or CBZ.
* Use of any investigational drug or participated in any clinical trial within the previous 2 months.
* Patient and/or his/her caregiver(s) unlikely to co-operate with the requirements of the study.
* If female, she was sexually active and of child-bearing potential and she did not use reliable contraception.
* Patients with non-epileptic attacks (syncopes, pseudoseizures).
* Previous poor compliance with anti-epileptic therapy.
* Need for rescue benzodiazepines more frequently than twice per week on average.
* Previous use of Eslicarbazepine acetate or participation in a clinical study with Eslicarbazepine acetate.
* Any other condition or circumstance that, in the opinion of the investigator, might compromise the patient's ability to comply with the clinical trial protocol (CTP).

At Visit 2, patient was not eligible for entry into the Eslicarbazepine acetate treatment phase if he/she fulfilled the following criteria:

* Inadequate compliance to concomitant AEDs during the baseline phase.
* Clinically relevant clinical laboratory test abnormalities at screening.
* Occurrence of any other condition or circumstance that, in the opinion of the investigator, might compromise the patient's ability to comply with the CTP.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2005-06; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica de Neurologie Pediatrica, Spitalul "Alexandru Obregia", Bucharest, Romania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 (2-6 Yrs) | Group 2 (7-11 Years) | Group 3 (12-17 Years)
Started | 15 | 9 | 11
Safety Population (SP) | 12 | 8 | 11
Pharmacokinetic Population (PKP) | 11 | 8 | 10
Efficacy Population (EP) | 11 | 8 | 10
Completed | 9 | 7 | 10
Not Completed | 6 | 2 | 1
Not completed — Withdrawal by Subject | 5 | 1 | 1
Not completed — Physician Decision | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1 (2-6 Yrs); Group 2 (7-11 Yrs); Group 3 (12-17 Yrs): Efficacy population (EP)
- Total: Total of all reporting groups
Arm/Group | Group 1 (2-6 Yrs) | Group 2 (7-11 Yrs) | Group 3 (12-17 Yrs) | Total
Number analyzed (Participants) | 11 | 8 | 10 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.1 (1.38) | 9.1 (1.55) | 14.5 (1.58) | 9.1 (4.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 3 | 17
  Male | 3 | 2 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Drug Concentration (Cmax) Post-dose
Time Frame: pre-dose, and ½, 1½, 3, 4½, 6 and 12 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1 (2-6 Yrs) | Group 2 (7-11 Yrs) | Group 3 (12-17 Yrs)
Number analyzed (Participants) | 11 | 8 | 10
ng/mL
  Dosage regimen 5 mg/kg/day | 6921 (1794) | 4820 (1693) | 6382 (1854)
  Dosage regimen 15 mg/kg/day | 16183 (2609) | 16395 (3680) | 17194 (3410)
  Dosage regimen 30 mg/kg/day | 29935 (4627) | 26890 (6944) | 32400 (6005)

2. Primary Outcome: Time of Occurrence of Cmax (Tmax).
Time Frame: pre-dose, and ½, 1½, 3, 4½, 6 and 12 hours post-dose
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Group 1 (2-6 Yrs) | Group 2 (7-11 Yrs) | Group 3 (12-17 Yrs)
Number analyzed (Participants) | 11 | 8 | 10
hours
  Dosage regimen 5 mg/kg/day | 1 (1) | 2 (1) | 2 (1)
  Dosage regimen 15 mg/kg/day | 2 (1) | 3 (1) | 2 (1)
  Dosage regimen 30 mg/kg/day | 1 (0) | 3 (1) | 3 (2)

3. Secondary Outcome: Percentage Change in Seizure Frequency During Each 4-week Treatment Period Compared to the Baseline Phase
Description: The efficacy variables were the percentage change in seizure frequency during each 4-week treatment period compared to the baseline phase.
  Seizures were recorded in the patient's diary during the baseline phase and during the following 4-week treatment periods.
  Seizure frequency for each patient was standardised to a frequency per 28 days period (i.e., mean daily frequency multiplied by 28). Changes in seizure frequency were analysed for each age group separately.
Time Frame: Baseline, end of 5 mg/kg/day treatment period (4 weeks), 15 mg/kg/day treatment period (4 weeks) and 30 mg/kg/day treatment period (4 weeks).
Measure: Median (95% Confidence Interval); unit: percent change
Arm/Group | Group 1 (2-6 Yrs) | Group 2 (7-11 Yrs) | Group 3 (12-17 Yrs)
Number analyzed (Participants) | 11 | 8 | 10
percent change
  5Dosage regimen 5 mg/kg/day | -28.2 [-60 to 13] | -11.7 [-20.0 to 278.2] | -17.1 [-56 to 30]
  Dosage regimen 15 mg/kg/day | -24.8 [-93 to -6] | 5.0 [-55.6 to 344.6] | -31.7 [-71 to 19]
  Dosage regimen 30 mg/kg/day | -40.6 [-86 to -4] | 12.2 [-100.0 to 166.7] | -43.1 [-77 to 21]

ADVERSE EVENTS:
Groups:
- Group 1 (2-6 Yrs); Group 2 (7-11 Yrs); Group 3 (12-17 Yrs): Safety population (SP)
Arm/Group | Group 1 (2-6 Yrs) | Group 2 (7-11 Yrs) | Group 3 (12-17 Yrs)
Serious Adverse Events (participants affected / at risk) | 2/12 | 1/8 | 0/11
Other Adverse Events (participants affected / at risk) | 9/12 | 7/8 | 7/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (2-6 Yrs) (N=12) | Group 2 (7-11 Yrs) (N=8) | Group 3 (12-17 Yrs) (N=11)
Seizures (Nervous system disorders) | 1 | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (2-6 Yrs) (N=12) | Group 2 (7-11 Yrs) (N=8) | Group 3 (12-17 Yrs) (N=11)
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Flu like symptoms (General disorders) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 5 | 3 | 0
Incoordination (Nervous system disorders) | 1 | 0 | 0
Psychomotor agitation (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 3 | 5
Aggressive behaviour (Psychiatric disorders) | 0 | 1 | 0
Interstitial pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2
Allergy to insect sting (Immune system disorders) | 1 | 0 | 0
Viral pharyngitis (Infections and infestations) | 1 | 0 | 0
Viral tonsillitis (Infections and infestations) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Drowsiness (Nervous system disorders) | 1 | 0 | 0
Acute pharyngitis (Infections and infestations) | 0 | 0 | 2
Inappetence (Metabolism and nutrition disorders) | 0 | 1 | 0
Equilibrium trouble (Nervous system disorders) | 0 | 0 | 1
Intention tremor (Nervous system disorders) | 0 | 2 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 2
Seizures (Nervous system disorders) | 1 | 1 | 0
Aggression aggravated (Psychiatric disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other